CLINICAL TRIAL: NCT02041377
Title: User Performance of the Karajishi Contour TS Blood Glucose Monitoring System
Brief Title: Evaluation of an Karajishi TS Investigational Blood Glucose Monitoring System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GCA-2013-002-01
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Results first posted 2015-02-16 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Monitoring System (Experimental): Subjects with diabetes used the Karajishi TS Investigational Blood Glucose Monitoring System with no training. The criteria for the intended use population:
  1. At least 60% of subjects will be younger than age 65
  2. At least 10% of subjects will have type 1 diabetes
  Interventions: Device: Karajishi TS Investigational Blood Glucose Monitoring System

INTERVENTIONS:
Device: Karajishi TS Investigational Blood Glucose Monitoring System — Subjects with diabetes performed self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the Karajishi TS Investigational Blood Glucose Monitoring System with no training. All BG results were compared to reference method results obtained from subject capillary plasma. Also, study staff tested subject venous blood and BG results were compared to reference method results obtained from subject venous plasma.

SUMMARY:
The purpose of this study was to determine if subjects who have diabetes can operate the Investigational Blood Glucose Monitoring System (BGMS) with no training and obtain valid glucose results.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 18 years of age and older
* People with type 1 or type 2 diabetes
* Able to speak, read, and understand English
* Willing to complete all study procedures

Exclusion Criteria:

* Hemophilia or any other bleeding disorder
* Pregnancy
* Physical, visual, or neurological impairments that would make the person unable to perform testing with the BGM
* Previously participated in a BG monitor study using the Karajishi TS BGMS (or used a Bayer Contour TS meter)
* Working for a medical laboratory, hospital, or other clinical setting that involves training on and clinical use of blood glucose monitors
* Working for a competitive medical device company, or having an immediate family member who works for such a company
* A condition which, in the opinion of the investigator or designee, would put the person or study conduct at risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Klaff, MD, Principal Investigator — Rainier Clinical Research Center; Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (2):
- United States (2):
  - AMCR Institute, Escondido, California
  - Rainier Clinical Research Center, Renton, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended Users of the Monitoring System: Subjects with diabetes used the Karajishi TS Investigational Blood Glucose Monitoring System with no training. The criteria for the intended use population:
  1. At least 60% of subjects will be younger than age 65
  2. At least 10% of subjects will have type 1 diabetes
  Karajishi TS Investigational Blood Glucose Monitoring System: Subjects with diabetes performed self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the Karajishi TS Investigational Blood Glucose Monitoring System with no training. All BG results were compared to reference method results obtained from subject capillary plasma. Also, study staff tested subject venous blood and BG results were compared to reference method results obtained from subject venous plasma.
Period: Overall Study
Arm/Group | Intended Users of the Monitoring System
Started | 134
Completed | 134
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 134
Age, Customized [Mean (Full Range); unit: years]
  Age of enrolled subjects | 53.8 [19 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71
  Male | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 121
  Unknown or Not Reported | 1
Race (NIH/OMB) [Number; unit: responses] — Subjects provided more than one choice for Race, therefore the apparent frequency total for Race was n=139.
  responses
    American Indian or Alaska Native | 3
    Asian | 8
    Native Hawaiian or Other Pacific Islander | 3
    Black or African American | 11
    White | 108
    More than one race | 5
    Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 134

OUTCOME MEASURES:

1. Primary Outcome: Number of Self-Test Fingerstick Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes self-tested fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS) with no training. BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI capillary plasma) and +/-15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 132 (134-2)Blood glucose results were analyzed. Lab reference replicates for one subject were discrepant and not evaluable per protocol. One subject had no fingerstick result.
Measure: Number; unit: Blood glucose results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 132
Blood glucose results | 127

2. Secondary Outcome: Number of Venous Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Study staff tested subject venous blood using an investigational Blood Glucose Monitoring System (BGMS). Venous BGMS results were compared with subject venous plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer venous plasma BG results were used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI venous plasma) and +/-15% (>=100 mg/dL YSI venous plasma).
Time Frame: 1 hour
Population: 131 (134-3) Blood glucose results were analyzed. Lab reference replicates for one subject were discrepant and not evaluable per protocol. Venipuncture was not successful for 2 subjects.
Measure: Number; unit: Blood glucose results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 131
Blood glucose results | 131

3. Secondary Outcome: Number of Blood Glucose (BG) Results From Alternative Site Testing (AST) Palm Blood Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method
Description: Subjects with diabetes self-tested Alternative Site (AST) palm blood using an investigational Blood Glucose Monitoring System (BGMS) with no training. BGMS AST palm results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI Analyzer BG results were used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI capillary plasma) and +/-15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 129 (134-5) Blood glucose results were analyzed. Lab reference replicates for one subject were discrepant and not evaluable per protocol. One subject had low blood sugar and AST result was not evaluable per protocol. One subject with low blood sugar did not attempt AST testing per protocol. No AST palm results were obtained for 2 subjects.
Measure: Number; unit: Blood glucose results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 129
Blood glucose results | 121

4. Secondary Outcome: Number of Subject Fingerstick Blood Glucose (BG) Results Within +/- 15 mg/dL (<100 mg/dL) and Within +/- 15% (>=100 mg/dL) of Laboratory Glucose Method When Obtained and Tested by Study Staff
Description: Study staff obtained and tested subject fingerstick blood using an investigational Blood Glucose Monitoring System (BGMS). BGMS results were compared with subject capillary plasma BG results obtained with a Yellow Springs Instrument (YSI) Analyzer. YSI capillary plasma results were used to calculate the number of BGMS results within +/-15 mg/dL (<100 mg/dL YSI capillary plasma) and +/-15% (>=100 mg/dL YSI capillary plasma).
Time Frame: 1 hour
Population: 133 (134-1) Blood glucose results were analyzed. Lab reference replicates for one subject were discrepant and not evaluable per protocol.
Measure: Number; unit: Blood glucose results
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 133
Blood glucose results | 131

5. Secondary Outcome: Number of Subject Responses That Strongly Agree or Agree or Are Neutral With Questionnaire Statements
Description: Staff obtained subject responses using short questionnaires to provide feedback on instructions for use and the basic operation of the BGMS. Subjects could respond Strongly Agree; Agree; Neutral; Disagree; or Strongly Disagree.
Time Frame: 1 hour
Measure: Number; unit: participants
Arm/Group | Intended Users of the Monitoring System
Number analyzed (Participants) | 134
participants
  I find it easy to do a blood test with this meter. | 132
  The meter display is easy to see and read. | 133
  It is easy to understand my test results. | 133
  I like the overall meter design. | 134
  I find the meter easy to use. | 132
  The instruction (User Guide) is easy to understand | 132
  Instructions clearly explain how to run a test. | 134
  Instructions clearly explain meter error messages. | 134

ADVERSE EVENTS:
Time Frame: 1 hour subject visit
Groups:
- Intended Users of the Monitoring System: Subjects with diabetes use the Karajishi TS Investigational Blood Glucose Monitoring System with no training. The criteria for the intended use population:
  1. At least 60% of subjects will be younger than age 65
  2. At least 10% of subjects will have type 1 diabetes
  Karajishi TS Investigational Blood Glucose Monitoring System: Subjects with diabetes perform self Blood Glucose (BG) tests with capillary fingerstick and palm blood using the Karajishi TS Investigational Blood Glucose Monitoring System with no training. All BG results are compared to reference method results obtained from subject capillary plasma. Also, study staff test subject venous blood and BG results are compared to reference method results obtained from subject venous plasma.
Arm/Group | Intended Users of the Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/134
Other Adverse Events (participants affected / at risk) | 2/134
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended Users of the Monitoring System (N=134)
Hypoglycemia (Endocrine disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days